CLINICAL TRIAL: NCT00628212
Title: A Phase II, Double-Blind, Placebo-Controlled, Monotherapy Study of MP-513 in Japanese Patients With Type 2 Diabetes Mellitus -Confirmative Study-
Brief Title: Efficacy and Safety Study of MP-513 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A4
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Teneligliptin 10 mg (Experimental): Teneligliptin 10 mg, orally, once daily
  Interventions: Drug: Teneligliptin 10mg
- Teneligliptin 20 mg (Experimental): Teneligliptin 20 mg, orally, once daily
  Interventions: Drug: Teneligliptin 20 mg
- Teneligliptin 40 mg (Experimental): Teneligliptin 40 mg, orally, once daily
  Interventions: Drug: Teneligliptin 40 mg
- Placebo (Placebo Comparator): Teneligliptin placebo-matching tablets, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teneligliptin 10mg
  Other Names: MP-513
  Arms: Teneligliptin 10 mg
Drug: Teneligliptin 20 mg
  Other Names: MP-513
  Arms: Teneligliptin 20 mg
Drug: Teneligliptin 40 mg
  Other Names: MP-513
  Arms: Teneligliptin 40 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety and to determine the appropriate dose for phase 3 confirmatory trial, of MP-513 (Teneligliptin) in patients with type 2 Diabetes based on the change of HbA1c and adverse events after 12 weeks administration once daily in multi-center, randomized, double-blind, placebo-controlled, parallel assignment manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 - 75 years old
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is 6.5 - 9.5%
* Patients who were not administered drugs prohibited for concomitant use within 12 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas failure, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients with Class III/IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Patients with serious diabetic complications
* Patients who are habitual excessive alcohol consumption.
* Patients with severe hepatic disorder or severe renal disorder.
* Pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, MD,PhD, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation; Tadashi Yoshida, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Takikawa-shi, Hokkaido, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Started | 80 | 84 | 79 | 81
Completed | 77 | 83 | 76 | 76
Not Completed | 3 | 1 | 3 | 5
Not completed — Adverse Event | 2 | 0 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg | Total
Number analyzed (Participants) | 80 | 84 | 79 | 81 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.6) | 57.7 (9.1) | 59.2 (9.5) | 57.5 (10.4) | 58.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 20 | 28 | 111
  Male | 51 | 50 | 59 | 53 | 213

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate.
Time Frame: 12 weeks
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization. Analysis based on last observation carried forward, where the last postbaseline double-blind observed value was carried forward and used for Week 12 where data was missing.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Number analyzed (Participants) | 80 | 84 | 79 | 81
Percent | 0.11 (0.05) | -0.77 (0.05) | -0.80 (0.05) | -0.91 (0.05)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: The change from Baseline in Fasting Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline Fasting Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Number analyzed (Participants) | 80 | 84 | 79 | 81
mg / dL | 2.8 (2.0) | -15.0 (2.0) | -14.1 (2.1) | -17.2 (2.0)

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in 2-hour Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline 2-hour Postprandial Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization.
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Number analyzed (Participants) | 80 | 84 | 79 | 81
mg / dL | 7.3 (4.5) | -43.3 (4.3) | -49.4 (4.5) | -51.3 (4.5)

4. Secondary Outcome: Change From Baseline in the Areas Under the Curve From 0 to 2 h (AUC0-2h) for Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in AUC0-2h for Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline AUC0-2h for Postprandial Plasma Glucose as a covariate.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg*h / dL
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Number analyzed (Participants) | 80 | 84 | 79 | 81
mg*h / dL | 5.897 (6.410) | -65.445 (6.141) | -73.211 (6.409) | -75.326 (6.422)

ADVERSE EVENTS:
Arm/Group | Placebo | Teneligliptin 10 mg | Teneligliptin 20 mg | Teneligliptin 40 mg
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/84 | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 44/80 | 50/84 | 40/79 | 46/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Teneligliptin 10 mg (N=84) | Teneligliptin 20 mg (N=79) | Teneligliptin 40 mg (N=81)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Teneligliptin 10 mg (N=84) | Teneligliptin 20 mg (N=79) | Teneligliptin 40 mg (N=81)
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 11 | 16 | 9 | 14
Onychomycosis (Infections and infestations) | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0
Tinea manuum (Infections and infestations) | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Neurogenic shock (Vascular disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Urticaria thermal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 2 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 6 | 1 | 4 | 3
Blood urine present (Investigations) | 1 | 4 | 2 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 4 | 4 | 2 | 2
Urobilin urine present (Investigations) | 0 | 0 | 1 | 0
Urine ketone body present (Investigations) | 1 | 3 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Deafness traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other